CLINICAL TRIAL: NCT01031485
Title: Bioactive Milk Peptides and Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valio Ltd (Industry)
Collaborators: University of Helsinki (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Valio-70
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Stage 1 Hypertension
Keywords: hypertension; blood pressure; milk peptides; bioactive peptides; randomized controlled trial
MeSH Terms: conditions — Hypertension | interventions — Phytosterols

ARMS (2):
- Spread with milk peptides and plant sterols (Active Comparator)
  Interventions: Dietary Supplement: Milk peptides and plant sterols
- Standard spread (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Milk peptides and plant sterols
  Arms: Spread with milk peptides and plant sterols
Other: Placebo
  Arms: Standard spread

SUMMARY:
The purpose of this study is to investigate the effects of bioactive milk peptides on blood pressure in mildly hypertensive subjects.

ELIGIBILITY:
Inclusion Criteria:

* age 30-60 years
* systolic blood pressure 140-160 mmHg and diastolic blood pressure 90-99 mmHg in office measurement
* apparently healthy

Exclusion Criteria:

* antihypertensive and lipid-lowering drugs
* unstable coronary artery disease, diabetes, malignant diseases, secondary hypertension
* BMI > 32 kg/m2
* milk allergy
* smoking
* alcohol abuse
* pregnancy, lactation
* simultaneous participation in other clinical trial

Ages: 30 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Valio Ltd, Helsinki, Uusimaa, Finland